CLINICAL TRIAL: NCT02433067
Title: Impact of Physical Activity Intervention on Myocardial Function in Patients With HER2 + Breast Cancer, During Treatment With Trastuzumab in Adjuvant
Brief Title: Physical Activity Intervention on Myocardial Function in Patients With HER2 + Breast Cancer
Acronym: CARDAPAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Franche-Comté (Other)
Collaborators: Ligue contre le cancer, France (Other); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Fabienne Mougin-Guillaume, Ph.D, University of Franche-Comté
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UFranche-Comte
Record Dates: First submitted 2015-04-14; First posted 2015-05-04 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention (Experimental): - Arm A "standard oncologic care coupled with physical activity intervention (3 times / week) " during 3 months
  Interventions: Other: Physical activity intervention
- Control group (Active Comparator): - Arm B (control group) "standard oncologic care"
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Physical activity intervention — Patients in arm A (interventional) will carry out a physical activity intervention during 3 months. Patients should perform an interval training program on cycle-ergometer during 3 sessions per week.
  Arms: Physical activity intervention
Other: Control Group — standard oncologic care
  Arms: Control group

SUMMARY:
Purpose of the study is to examine the effects of 3 months of physical activity intervention on myocardial function (Left ventricular ejection fraction) in patients with HER2+ breast cancer

DETAILED DESCRIPTION:
Primary objective: To evaluate in patients with HER2 + breast cancer, treated only by trastuzumab, the impact of three months individualized physical activity intervention (55 minutes, 3 times per week) on left ventricular ejection fraction (LVEF).

Secondary objectives: To evaluate the impact of physical activity intervention on body composition, muscle function, metabolic, hormonal and inflammatory responses, pain, fatigue and quality of life.

This study examines patients aged 18 to 85 years, diagnosed with early breast cancer with HER2 overexpression confirmed histologically and eligible to receive treatment with trastuzumab (adjuvant).

This study includes 3 assessments phases: baseline (T0), 3 months (T3) and 6 months (T6) for both arms.

The programme is organised as follows: Arm A "standard oncologic care coupled with physical activity intervention (3 times / week) " for 3 months ; Arm B (control group) "standard oncologic care".

Between T3 and T6, volontary physical activity level will follow by actimetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years
* First breast cancer HER2 + histologically confirmed,
* WHO grade Performance Index ≤1
* Normal renal function (creatinine clearance ≥ 60 ml min-1)
* Normal heart function with LVEF ≥ 50%
* Normal liver function (AST and ALT normal)
* Physical activity certificate issued by a cardiologist or an oncologist,
* Active contraception or postmenopausal

Exclusion Criteria:

* Patients aged under 18 and over 85
* Patients having no breast cancer HER2+
* Patients with metastases
* Heart failure (LVEF ≤50%) and respiratory (O2 saturation ≤ 92%),
* Autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis)
* Symptomatic osteoarthritis,
* Cardiovascular diseases (angina or uncontrolled high blood pressure) or heart-lung (chronic obstructive pulmonary disease)
* Patients suffering from malnutrition (Body Mass Index (BMI) <18 kg m-2) or weight loss of over 10% during the last 3 months,
* Patients with psychiatric or cognitive disorders deemed unsuitable for a sporting activity
* Pregnant or lactating Patients.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-04; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | The Left Ventricular Ejection Fraction (LVEF) will be evaluated baseline (T0), and 6 months (T6), to see if there is a significant change
  evaluated with echocardiography

SECONDARY OUTCOMES:
Weight and volume of left and right ventricular | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with echocardiography
Body composition | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated byimpedance and with tape measure and pliers of Harpenden
Metabolic responses | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with enzyme-linked immunosorbent assay (ELISA)
Maximal voluntary quadriceps | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with chair quadriceps with strain gauge
score of Quality of life | Baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with questionnaire
score of Pain | Baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with questionnaire
Fatigue | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with questionnaire
Level of physical activity | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with questionnaire
Pulmonary function (at rest and during exercise) | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with respiratory functional test and maximal exercise test
hormonal responses | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with enzyme-linked immunosorbent assay (ELISA)
inflammatory responses | baseline (T0), 3 months (T3) and 6 months (T6)
  evaluated with enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Meneveau, Principal Investigator — University Hospital of Besançon
Locations (1):
- University Hospital, Besançon, Doubs, France

REFERENCES:
- [Derived] Jacquinot Q, Ennequin G, Falcoz A, Sawyer D, Meneveau N, Mougin F. Exercise training decreases Neuregulin-1 concentrations in HER2-positive breast cancer patients undergoing adjuvant trastuzumab: the CARDAPAC study. Breast Cancer Res Treat. 2026 Feb 4;215(3):69. doi: 10.1007/s10549-026-07903-x. PMID 41636910
- [Derived] Jacquinot Q, Meneveau N, Falcoz A, Bouhaddi M, Roux P, Degano B, Chatot M, Curtit E, Mansi L, Paillard MJ, Bazan F, Chaigneau L, Dobi E, Meynard G, Vernerey D, Pivot X, Mougin F. Cardiotoxicity is mitigated after a supervised exercise program in HER2-positive breast cancer undergoing adjuvant trastuzumab. Front Cardiovasc Med. 2022 Sep 23;9:1000846. doi: 10.3389/fcvm.2022.1000846. eCollection 2022. PMID 36211552
- [Derived] Jacquinot Q, Meneveau N, Chatot M, Bonnetain F, Degano B, Bouhaddi M, Dumoulin G, Vernerey D, Pivot X, Mougin F. A phase 2 randomized trial to evaluate the impact of a supervised exercise program on cardiotoxicity at 3 months in patients with HER2 overexpressing breast cancer undergoing adjuvant treatment by trastuzumab: design of the CARDAPAC study. BMC Cancer. 2017 Jun 19;17(1):425. doi: 10.1186/s12885-017-3420-4. PMID 28629338